CLINICAL TRIAL: NCT07311694
Title: A Phase III, Randomized, Open-Label, Multicenter Study Comparing HRS-4357 With Novel Androgen Receptor Pathway Inhibitors in Patients With Progressive, PSMA-Positive Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase III Study Comparing HRS-4357 With Novel Androgen Receptor Pathway Inhibitors in Patients With Progressive, PSMA-Positive Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4357-301
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: PSMA-Positive Progressive Metastatic Castration-Resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-4357 injection (Experimental)
  Interventions: Drug: HRS-4357 injection
- Enzalutamide Soft Capsules / Abiraterone Acetate Tablets+ Prednisone Acetate Tablets (Active Comparator)
  Interventions: Drug: Enzalutamide；Abiraterone

INTERVENTIONS:
Drug: HRS-4357 injection — HRS-4357 injection are administered each time, with dosing for 4 to 6 cycles
  Arms: HRS-4357 injection
Drug: Enzalutamide；Abiraterone — ARPI (investigator's choice of any of the following agents, with the requirement that the agent has not been used previously):
  * Enzalutamide 160 mg orally once daily (qd)
  * Abiraterone 1000 mg orally once daily (qd) + Prednisone 5 mg orally twice daily (bid)
  Arms: Enzalutamide Soft Capsules / Abiraterone Acetate Tablets+ Prednisone Acetate Tablets

SUMMARY:
This study is a randomized, open-label, controlled, multicenter phase III clinical trial, which plans to randomly enroll 370 subjects with advanced metastatic castration-resistant prostate cancer (mCRPC). The efficacy of HRS-4357 versus novel androgen receptor pathway inhibitors (ARPI) in the treatment of PSMA-positive advanced metastatic castration-resistant prostate cancer (mCRPC) will be evaluated based on radiographic progression-free survival (rPFS) assessed by the BIRC.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to participate in this clinical trial, understand the study procedures, and be able to sign the informed consent form in writing;
2. Male, aged ≥ 18 years;
3. ECOG performance status score of 0-1;
4. Expected survival time of no less than 6 months;
5. Prostate adenocarcinoma confirmed by histology and/or cytology, and diagnosed as mCRPC (metastatic castration-resistant prostate cancer) with reference to current clinical guidelines;
6. Presence of at least one metastatic lesion confirmed by imaging examinations (CT/MRI and/or bone scan) within 4 weeks before randomization;
7. Confirmation of at least one PSMA-positive lesion and no PSMA-negative lesions by PSMA PET/CT;
8. Serum testosterone at castration level (< 50 ng/dl or < 1.7 nmol/L) at the screening visit; continuous luteinizing hormone-releasing hormone analog (LHRHA) therapy (medical castration) or previous bilateral orchiectomy (surgical castration); subjects who have not undergone bilateral orchiectomy must plan to maintain effective LHRHA therapy throughout the study period;
9. Previous treatment with second-generation ARPIs, with only one episode of disease progression during treatment; and assessed by the investigator as suitable for switching to another ARPI (suitable for receiving abiraterone or enzalutamide);
10. Disease progression at the time of enrollment. Disease progression is defined as the occurrence of at least one of the following while the subject's serum testosterone is at a stable castration level: ① PSA progression: PSA value > 1 ng/mL, with two consecutive increases in PSA at intervals of at least 1 week; ② Radiographic progression: occurrence of clearly new lesions; appearance of 2 or more new bone lesions on bone scan; lesion progression indicated by CT or MRI (per RECIST v1.1);

Exclusion Criteria:

1. Received any of the following treatments before randomization:

   1. Any radionuclide therapy or hemi-body radiotherapy within 6 months.
   2. Any PSMA-targeted radiopharmaceutical therapy.
   3. Surgery, radiotherapy, or any local therapy within 4 weeks.
   4. Any other investigational drug intervention within 4 weeks.
2. Known hypersensitivity to the components of the study drug or its analogs.
3. History of malignancy (other than prostate cancer) within 5 years before randomization that is expected to alter life expectancy or may interfere with disease assessment, excluding cured malignancies with low risk of metastasis and mortality (5-year survival rate > 90%), such as non-metastatic basal cell carcinoma of the skin, superficial squamous cell carcinoma of the skin, and low-grade superficial bladder cancer.
4. Occurrence of severe infection (CTCAE > Grade 2) within 4 weeks before randomization.
5. Failure to recover from adverse events of previous treatments (NCI-CTCAE Version 5.0 Grade > 1) before randomization, as judged by the investigator.
6. Presence of poorly controlled clinical cardiac symptoms or cardiac diseases.
7. History of physical or psychiatric illnesses/conditions that may interfere with the study objectives and assessments (including epilepsy and dementia).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
radiographic progression-free survival (rPFS) assessed by the BIRC. | From Baseline to primary completion date, about 24 months

SECONDARY OUTCOMES:
OS | From Baseline to primary completion date, about 24 months
rPFS（Investigator-Assessed） | From Baseline to primary completion date, about 24 months
ORR （Investigator-Assessed and BIRC-Assessed） | From Baseline to primary completion date, about 24 months
DCR（Investigator-Assessed and BIRC-Assessed） | From Baseline to primary completion date, about 24 months
DOR（Investigator-Assessed and BIRC-Assessed） | From Baseline to primary completion date, about 24 months
PSA50 Response Rate | From Baseline to primary completion date, about 24 months
Time to PSA Progression | From Baseline to primary completion date, about 24 months
Changes from baseline in scores of the EQ-5D-5L | From Baseline to primary completion date, about 24 months
Changes from baseline in scores of the Functional FACT-P | From Baseline to primary completion date, about 24 months
Changes from baseline in scores of the BPI-SF | From Baseline to primary completion date, about 24 months
Assessment of the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From Baseline to primary completion date, about 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided